CLINICAL TRIAL: NCT03069469
Title: A Multicenter Phase 1/2, Open-Label Study of DCC-3014 to Assess the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics in Patients With Advanced Tumors and Tenosynovial Giant Cell Tumor
Brief Title: Study of Vimseltinib (DCC-3014) in Patients With Advanced Tumors and Tenosynovial Giant Cell Tumor
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCC-3014-01-001; 2024-514933-39-00 (EU CTIS Number)
Record Dates: First submitted 2017-02-20; First posted 2017-03-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Neoplasm; Pigmented Villonodular Synovitis; Giant Cell Tumor of Tendon Sheath; Tenosynovial Giant Cell Tumor; Tenosynovial Giant Cell Tumor, Diffuse
Keywords: TGCT; DTGCT; PVNS
MeSH Terms: conditions — Synovitis, Pigmented Villonodular; Giant Cell Tumor of Tendon Sheath

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Treatment (Other): Dose Escalation Phase: Increasing doses of vimseltinib beginning at 10 milligram (mg) once daily (QD) for 28 day cycles until disease progression or unacceptable toxicity.
  Expansion Phase: Dosing of different patient cohorts at the dose level determined from the Dose Escalation Phase of the study.
  Interventions: Drug: Vimseltinib

INTERVENTIONS:
Drug: Vimseltinib — Colony-stimulating factor 1 receptor (CSF1R) inhibitor
  Other Names: DCC-3014

SUMMARY:
This is a multicenter, open-label Phase 1/2 study of vimseltinib in patients with malignant solid tumors and tenosynovial giant cell tumor (TGCT). There will be 2 distinct parts in this study: Dose Escalation (Phase 1) and Expansion (Phase 2). Phase 1 will enroll both malignant solid tumor and TGCT patients. Phase 2 will comprise two cohorts (Cohort A and Cohort B) and will only enroll TGCT patients.

ELIGIBILITY:
Inclusion Criteria

Dose Escalation Phase:

1. Patients ≥18 years of age
2. Patients must have:

   1. advanced malignant solid tumors; or
   2. symptomatic TGCT for which surgical resection is not an option (tumor biopsy to confirm diagnosis required if no histology/pathology available at screening)
3. Malignant solid tumor patients only: Able to provide a tumor tissue sample
4. Must have 1 measurable lesion according to RECIST Version 1.1
5. Malignant solid tumor patients only: Must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
6. Adequate organ and bone marrow function
7. If a female of childbearing potential, must have a negative pregnancy test prior to enrollment and agree to follow the contraception requirements.
8. Must provide signed consent to participate in the study and is willing to comply with study-specific procedures.

Expansion Phase (Cohorts A and B)

1. Patients ≥18 years of age
2. Patients must have symptomatic TGCT for which surgical resection is not an option (tumor biopsy to confirm diagnosis required if no histology/pathology available at screening)

   a) Expansion Cohort B: patients must have prior systemic treatment with anti-CSF1 or anti-CSF1R therapy, with the exception of imatinib or nilotinib
3. Adequate organ and bone marrow function
4. Must have at least 1 measurable lesion according to RECIST Version 1.1
5. If a female of childbearing potential, must have a negative pregnancy test prior to enrollment and agree to follow the contraception requirements.
6. Must provide signed consent to participate in the study and is willing to comply with study-specific procedures.

Exclusion Criteria

Dose Escalation Phase:

1. Received anticancer therapy or therapy for TGCT, including investigational therapy, within 2 weeks or 28 days for therapies with half-life (t1/2) longer than 3 days prior to the administration of study drug.
2. Unresolved toxicity (Grade >1 or baseline) from previous anticancer therapy or TGCT therapy, excluding alopecia.
3. Known active central nervous system (CNS) metastases.
4. History or presence of clinically relevant cardiovascular abnormalities.
5. Systemic arterial or venous thrombotic or embolic events.
6. QT interval corrected by Fridericia's formula (QTcF) >450 ms in males or >470 ms in females or history of long QT syndrome.
7. Left ventricular ejection fraction (LVEF) <50%.
8. Concurrent treatment with proton-pump inhibitor(s).
9. Major surgery within 2 weeks of the first dose of study drug.
10. Malabsorption syndrome or other illness that could affect oral absorption.
11. Known human immunodeficiency virus, active hepatitis B, active hepatitis C, or active mycobacterium tuberculosis infection.
12. If female, the patient is pregnant or lactating.
13. Known allergy or hypersensitivity to any component of the study drug.
14. Any other clinically significant comorbidities.

Expansion Phase (Cohorts A and B)

1. Expansion Cohort A: received systemic therapy targeting CSF1 or CSF1R; previous therapy with imatinib and nilotinib is allowed.
2. Expansion Cohort B: discontinued systemic therapy targeting anti-CSF1 or anti-CSF1R due to drug-induced liver injury.
3. Treatment with therapy for TGCT, including investigational therapy, within 2 weeks or 28 days for therapies with a t1/2 longer than 3 days prior to the administration of the study drug.
4. Known metastatic TGCT or other active cancer that requires concurrent treatment.
5. QT interval corrected by Fridericia's formula (QTcF) >450 ms in males or >470 ms in females or history of long QT syndrome.
6. Left ventricular ejection fraction (LVEF) <55%.
7. Concurrent treatment with proton-pump inhibitor(s).
8. Major surgery within 2 weeks of the first dose of study drug.
9. Any clinically significant comorbidities
10. Malabsorption syndrome or other illness that could affect oral absorption.
11. Known human immunodeficiency virus (HIV), active or chronic hepatitis B, active or chronic hepatitis C, or active mycobacterium tuberculosis infection.
12. If female, the patient is pregnant or lactating.
13. Known allergy or hypersensitivity to any component of the study drug.
14. Contraindication for MRI
15. Active liver or biliary disease, including evidence of fatty liver, nonalcoholic steatohepatitis (NASH), or cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Day 1 - Day 28 of Cycle 1 for each dose level tested
  Determine the maximum tolerated dose.
Number of Patients with Dose-Limiting Toxicities (DLTs) | Day 1- Day 28 of Cycle 1 for each dose level tested
  Identify the number of patients with DLTs for each dose level tested.
Time to maximum observed concentration of Vimseltinib | Cycle 1 Day 1 and Day 8, and Cycle 2 Day 1 (pre-dose and at multiple time points (up to 8 hours) post-dose)
  Measure the time to maximum plasma concentration of vimseltinib in patients.
Maximum observed concentration of Vimseltinib | Cycle 1 Day 1 and Day 8, and Cycle 2 Day 1 (pre-dose and at multiple time points (up to 8 hours) post-dose)
  Measure the maximum observed concentration of vimseltinib in patients.
Trough observed concentration of Vimseltinib | Cycle 1 Day 1 and Day 8, and Cycle 2 Day 1 (pre-dose and at multiple time points (up to 8 hours) post-dose)
  Measure the observed trough concentration of vimseltinib in patients.
Area under the concentration-time curve (AUC) of Vimseltinib | Cycle 1 Day 1 and Day 8, and Cycle 2 Day 1 (pre-dose and at multiple time points (up to 8 hours) post-dose)
  Measure the AUC of vimseltinib.
Half life of Vimseltinib | Cycle 1 Day 1 and Day 8, and Cycle 2 Day 1 (pre-dose and at multiple time points (up to 8 hours) post-dose)
  Measure half life of vimseltinib in patients.
Objective response rate (ORR= complete response [CR]+partial response [PR]) (Expansion Phase only) | At Week 25 (Cycle 7, Day 1)
  Assessed by central read using Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.
Duration of response rate (DOR) (Expansion Phase only) | Date from PR or CR to disease progression or death (Estimated up to 24 months)
  Measure time from partial response (PR) or complete response (CR) to disease progression or death.

SECONDARY OUTCOMES:
Response rate (Expansion Phase only) | At Week 25 (Cycle 7, Day 1)
  Assessed by central read using tumor volume score and modified RECIST (mRECIST) Version 1.1
Range of Motion (ROM) (Expansion Phase only) | Baseline to Week 25 (Cycle 7, Day 1)
  Measure mean change from baseline in relative ROM
Brief Pain Inventory (BPI) Worst Pain Numeric Rating Scale (NRS) Score (Expansion Phase only) | Baseline to Week 25 (Cycle 7, Day 1)
  Proportion of responders based on Brief Pain Inventory (BPI) worst pain numeric rating scale (NRS) and narcotic analgesic use by Brief Pain Inventory-30 (BPI-30)
Patient-reported Outcomes Measurement Information System (PROMIS) Physical Function Score (Expansion Phase only) | Baseline to Week 25 (Cycle 7, Day 1)
  Analysis of patient reported outcomes based upon the patient-reported outcomes measurement information system (PROMIS) physical function questionnaire
Worst Stiffness Numeric Rating Scale (NRS) Score (Expansion Phase only) | Baseline to Week 25 (Cycle 7, Day 1)
  Analysis of patient reported outcomes based upon the Worst Stiffness Numeric Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Maitreyi Sharma, MD, Study Director — Deciphera Pharmaceuticals, LLC
Locations (24):
- United States (9):
  - Stanford Cancer Institute, Palo Alto, California
  - University of Colorado - Denver, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Dana Farber, Boston, Massachusetts
  - MSKCC, New York, New York
  - OHSU, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Peter MacCallum Cancer Centre, Melbourne, Australia
- Canada (2):
  - McGill University Health Centre, Montreal, Quebec
  - Princess Margaret Cancer Center, Toronto
- France (2):
  - Centre Leon Berard, Lyon
  - Gustave Roussy Cancer Campus Grand Paris, Paris
- Italy (4):
  - IRCCS Istituto Ortopedico Rizzoli, Bologna
  - Fondazione IRCCS Istituto Nazionale Dei Tumori, Milan
  - Istituto Nazionale dei Tumori, Milan
  - Regina Elena National Cancer Institute, Rome
- Leiden University Medical Center, Leiden, Netherlands
- M. Sklodowska-Curie Memorial Cancer Center, Warsaw, Poland
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen del Rocío, Sevilla, Seville
- University College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No